CLINICAL TRIAL: NCT04662580
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation, and Dose-Expansion Study to Evaluate the Safety, Pharmacokinetics, and Anti-Tumor Activity of ARX517 as Monotherapy and in Combination With Androgen Receptor Pathway Inhibitors in Subjects With Metastatic Prostate Cancer
Brief Title: ARX517/JNJ-95298177 as Monotherapy or Combination Therapy in Subjects With Metastatic Prostate Cancer
Acronym: ARX517
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARX517-2011; ARX517-2011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-09-12; First posted 2020-12-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Prostate Cancer
Keywords: ADC; Antibody drug conjugate; Prostate neoplasia; Metastatic castration-resistant prostate cancer; PSMA; Prostate specific membrane antigen; PSMA ADC; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Intervention Model Description: This study has dose-escalation (Phase 1a) and dose-expansion (Phase 1b) stages to identify the maximum tolerated dose (MTD) and/or recommended development doses (RDDs) of ARX517. The initial treatment regimen is by weight-based infusion at an interval of every 3 weeks. In the Phase 1b dose expansion stage, the Sponsor will evaluate cohorts with alternative dose regimens to determine RDD(s). The term "alternative dose regimen" refers to any monotherapy treatment regimen where ARX517 is not given at a fixed interval of every 3 weeks.
  In the Phase 1b dose expansion stage, the Sponsor will also evaluate the safety and preliminary anti-tumor activity of ARX517 in combination with ARPIs (apalutamide or abiraterone acetate plus prednisone). ARPIs will be administered at the approved doses per product information. The starting dose of ARX517 to be given in combination with ARPIs will be determined by data emerging from the monotherapy dose expansion stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ARX517 (Experimental): ARX517 will be administered via intravenous (IV) infusion, with the initial treatment regimen by weight-based infusion at an interval of every 3 weeks. Other treatment regimen may be explored.
  Interventions: Drug: ARX517
- ARX517+Apalutamide (Experimental): ARX517 and apalutamide
  Interventions: Drug: ARX517; Drug: Apalutamide
- ARX517+AAP (Experimental): ARX517 and abiraterone acetate plus prednisone(AAP)
  Interventions: Drug: ARX517; Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: ARX517 — ARX517 is an ADC consisting of a humanized anti-PSMA monoclonal antibody (mAb) (IgG1κ) covalently conjugated to two (2) proprietary microtubule-disrupting toxins referred to as AS269.
Drug: Apalutamide — Oral tablet and will be given once daily by mouth.
  Arms: ARX517+Apalutamide
Drug: Abiraterone acetate — Oral tablet and will be given once daily by mouth.
  Arms: ARX517+AAP
Drug: Prednisone — Oral tablet and will be given once daily in metastatic castration-sensitive prostate cancer( mCSPC) and twice daily in metastatic castration-resistant prostate cancer (mCRPC) cohort by mouth.
  Arms: ARX517+AAP

SUMMARY:
This is a phase 1 study to assess the safety and tolerability of ARX517 as monotherapy or combination therapy in adult subjects with metastatic prostate cancer (mPC).

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, multicenter, open-label, dose-escalation and dose-expansion study to evaluate the safety, PK, pharmacodynamic (PDy), and preliminary anti-tumor activity of ARX517 alone, or in combination with androgen receptor pathway inhibitors (ARPIs), in adult subjects with metastatic prostate cancer .

ELIGIBILITY:
Key Inclusion Criteria:

* Male and ≥18 years at the time of providing written informed consent.
* Histologically confirmed prostate adenocarcinoma.
* For subjects who have not undergone an orchiectomy, must be undergoing treatment with a luteinizing hormone-releasing hormone (LHRH) agonist or antagonist and must agree to continue such therapy while on study treatment. Subjects enrolled to mCRPC cohorts must have serum testosterone levels of ≤50ng/dL (1.73nM at Screening).
* Must receive prior treatment(s) as defined in the protocol for each cohort
* Documented evidence of disease progression on or after the most-recent prior regimen for mCRPC cohorts
* mCSPC combination cohorts: High volume metastatic disease documented by CT/MRI and/or 99mTC bone scan (for bone lesions)
* Adequate blood counts
* Must have at least 1 PSMA-positive metastatic lesion and no measurable PSMA-negative lesions by local assessment for alternative dosing regimen and combination cohorts.

Key Exclusion Criteria

* Receipt of chemotherapy within 21 days prior to enrollment; hormonal therapy (not including LHRH analogs) within 7 days prior to enrollment; palliative radiation therapy within 7 days prior to enrollment; or any other anticancer therapy within 21 days prior to enrollment or other therapy for monotherapy cohorts
* Receipt of more than 1 prior taxane regimen or non-taxane chemotherapy for prostate cancer for alternative dose regimen and mCRPC combination cohorts
* Receipt prior apalutamide, enzalutamide, or darolutamide, or AAP for mCRPC combination cohorts
* Receipt any prior chemotherapy or prior ARPI, and must be greater than 90 days of ADT prior to enrollment for mCSPC combination cohorts
* Use of chronic systemic glucocorticoids equivalent to > 10 mg prednisone daily. Note: short-term administration of systemic corticosteroids > 10 mg prednisone equivalent (e.g., for allergic reactions or management of immune- or infusion-related AEs) is allowed.
* Symptomatic and/or untreated central nervous system (CNS) metastases. Patients with asymptomatic, untreated CNS metastases are eligible provided they have been clinically stable (neurologically stable and not requiring steroids for at least 28 days prior to enrollment).
* History of any invasive malignancy (other than primary) within the previous 2 years prior to the enrollment date that requires active therapy or is at high risk of recurrence in the opinion of the investigator.
* Marked baseline prolongation of QT/QT interval corrected for heart rate (QTc), e.g., a triplicate-average QTc interval > 480 milliseconds (CTCAE Grade 2) using Fridericia's QT correction formula at any time within 28 days before enrollment, ongoing history of CTCAE Grade ≥2 QTc at enrollment, or anticipated need to perform repeat ECG evaluations to satisfy re-treatment criteria.
* Prior history of interstitial lung disease, pneumonitis, or other clinically significant lung disease within 12 months prior to enrollment date.
* Clinically significant ocular findings by a qualified ophthalmologist or optometrist including active ocular infections or chronic corneal disorders unless approved by the Medical Monitor.
* Peripheral neuropathy Grade ≥ 2 within 28 days prior to enrollment.
* For combination cohorts with apalutamide: no prior history of seizure or condition that may predispose to seizure (including but not limited to prior cerebrovascular accident, TIA or loss of consciousness within the last 12 months, brain AVM, brain metastases).
* 24-hour urine protein > 1g/24h

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants only
Enrollment: 183 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Assess incidence of adverse events | 1.5 Years
  Incidence and severity of adverse events or serious adverse events of ARX517 alone or in combination with ARPIs will be assessed to determine the safety and tolerability of the treatment using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5 (CTCAE).

SECONDARY OUTCOMES:
Area under the serum concentration-time curve (AUC) for ARX517 alone or in combination with ARPIs | 3 Year
  Pharmacokinetic parameter area under the serum concentration-time curve (AUC) will be analyzed through different analytes such as ADC, total antibody, and pAF-AS269
Maximum serum concentration (Cmax) for ARX517 alone or in combination with ARPIs | 3 Year
  Pharmacokinetic parameter maximum serum concentration (Cmax) will be analyzed through different analytes such as, ADC, total antibody, and pAF-AS269
Trough concentration (Ctrough) for ARX517 alone or in combination with ARPIs | 3 Year
  Pharmacokinetic parameter trough concentration (Ctrough) will be analyzed through different analytes such as, ADC, total antibody, and pAF-AS269
Incidence of ADA against ARX517 alone or in combination with ARPIs | 3 year
  To assess the incidence of anti-drug antibodies (ADA) against ARX517 at selected timepoints
Overall survival (OS) | 3 year
  Overall survival (OS) is defined as the time from first dose of study therapy to the date of death (any cause). Subjects who are alive will be censored at the last known time that the subject was alive.
Assess changes in serum prostate specific antigen (PSA) levels | 3 year
  Proportion of subjects who show a confirmed reduction of 30%, 50%,and 90% from baseline in serum prostate specific antigen (PSA) levels (PSA30, PSA50, PSA 90)
Progression-free survival (PFS) | 3 year
  PFS is defined as the time between date of first dose of study therapy and date of progression or death, whichever occurs first, will be computed for response evaluable subjects. Subjects will be censored at time of subsequent therapy

OTHER OUTCOMES:
Evaluate of biomarkers | 3 years
  To evaluate exploratory blood based biomarkers related to study drug response
Evaluate PSMA expression | 3 years
  To evaluate relationship of PSMA expression and anti-tumor activity
Assess changes in Brief Pain Inventory-Short Form (BPI-SF) | 3 year
  A Brief Pain Inventory questionnaire will be utilized to assess subject quality of life. Higher scores mean a worse outcome
Assess changes in Functional Assessment of Cancer Therapy for Patients with Prostate Cancer (FACIT-P) | 3 year
  FACT-P questionnaire will be utilized to assess subject quality of life. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (12):
- United States (12):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles School of Medicine, Los Angeles, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University St. Louis School Medicine Siteman Cancer Center, St Louis, Missouri
  - GU Research Network, Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Skidmore LK, Mills D, Kim JY, Knudsen NA, Nelson JD, Pal M, Wang J, Gc K, Gray MJ, Barkho W, Nagaraja Shastri P, Ramprasad MP, Tian F, O'Connor D, Buechler YJ, Zhang SS. Preclinical Characterization of ARX517, a Site-Specific Stable PSMA-Targeted Antibody-Drug Conjugate for the Treatment of Metastatic Castration-Resistant Prostate Cancer. Mol Cancer Ther. 2024 Dec 3;23(12):1842-1853. doi: 10.1158/1535-7163.MCT-23-0927. PMID 39172730